CLINICAL TRIAL: NCT04705428
Title: Preventive Therapy of White Spot Lesions Using Different Remineralizing Agents in Children From 3 to 12 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Francisco Guinot-Jimeno, Jefe departamento de odontopedaitria, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UIC-ODP-WHITE SPOT
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: intervention group 1 (Experimental): Professional hygiene will be carried out with the application of fluoride varnish (Duraphat) and the use of fluoride paste according to the age will be recommended for oral hygiene at home.
  Interventions: Other: FLUORINE VARNISH
- Group II: intervention group 2 (Experimental): Professional hygiene will be carried out with the application of fluorine varnish (Tiefenfluoride) and the use of fluoride paste according to the age will be recommended for oral hygiene at home.
  Interventions: Other: FLUORINE VARNISH
- Group III: intervention group 3 (Experimental): Professional hygiene will be carried out with the application of fluorine varnish (Fluor Protector S) and the use of fluoride paste according to the age will be recommended for oral hygiene at home.
  Interventions: Other: FLUORINE VARNISH

INTERVENTIONS:
Other: FLUORINE VARNISH — Participants in all groups will receive written oral hygiene and oral prophylaxis instructions. All groups will receive the application of fluorine varnish every 3 months.
  The application of fluoride in the three groups will be done as follows:
  -Drying of the teeth, placement of the fluorine varnish on the teeth by quadrants. The varnish will be left to dry for a few seconds according to the manufacturer's instructions. Children in all groups will be asked to avoid brushing and flossing for one day after applying fluoride. They will be instructed to avoid hard food and hot drinks for 4 hours. Children and parents will be instructed on how to care for their teeth at home: brush teeth with conventional toothpaste containing 1000 ppm sodium fluoride, for 3 minutes without rinsing.
  In the following reviews (3 and 6 months) the effectiveness of the treatments will be evaluated by visual examination, tactile examination, fluorescence and photography.
  Other Names: 3 MONTHS; 6 MONTHS

SUMMARY:
Compare by clinical observation, photographs and fluorescence the efficacy of sodium fluoride, silanofluoride and thiefenfluoride in treating white spots.

DETAILED DESCRIPTION:
This in vivo study will be a randomized experimental clinical trial to be carried out in the Department of Pediatric Dentistry of the International University of Catalonia. Patients between the ages of 3 and 12, who attend the dental university clinic of the International University of Catalonia, will be part of the study.

Parents or legal guardians will be informed of the treatment procedure with a patient information sheet and informed consent will be given. Once signed, the patient will be assigned to one of the 3 study groups.

Accepting an alpha risk of 5% and with a power of 80% in a bilateral contrast, 15 subjects in each group are required to detect a minimum difference of 4 points between two groups, assuming that there are 3 groups and a standard deviation of 4.9. a follow- up loss rate of 10% has been estimated. The total number of children will be 45 by 15 for each group.

In order to analyze the degree of agreement of one examiner, 15 children will be evaluated twice, with a separation of one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients born between 2008 and 2017 of both sexes
* Patients with the active white spot lesions on vesicular and buccal surfaces of the incisors and molars of different sizes and with or without sensitivity to external stimuli
* Patients with white spot lesions that correspond to codifications of 0 to 2 of the ICDAS criteria.

Exclusion Criteria:

* Patients with mental disabilities or systemic diseases
* Patients with previously restored teeth
* Patients with clinical symptoms of irreversible pulpitis, allergy to fluoride and copper

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
visual examination, | 6 MONTHS
  Clinical examination, using ICDAS criteria for the visual diagnosis of caries. The visual inspection will be carried out using the ICDAS criteria. Selected sites will be examined with direct visualization under light illumination and a three-in-one air syringe, without probing. Wet teeth will be evaluated first, and then dried after 5 s. Visual examination will be coded as follows: (0) healthy tooth surfaces, with no evidence of caries after prolonged air drying (5 s); (1) white or brown stain visible on dry enamel; (2) white or brown stain visible on wet enamel. Teeth with codes from 0 to 2 will be included in the study.
tactile examination | 6 MONTHS
  Tactile examination. An exploratory probe will be used by moving it over the examination surfaces without applying pressure. The data will be recorded as follows: 1. Smooth surface, 2 Rough surface, based on a modification of the criteria of Ekstrand et al.
fluorescence | 6 MONTHS
  Using the quantitative light fluorescence method using a VistaProof device (Dürr Dental), the use of which significantly improves the quality of the diagnoses. The results will be evaluated by recording the indications of fluorescence intensity before and after treatment. The fluorescence chamber will be positioned up, parallel to the buccal / buccal surface. The software (DBSWIN, Dürr Dental) will digitize the video signal to create buccal / buccal surface images of 720 × 576 pixels with 3 × 8 bit RGB channel intensities and a resolution of 72 pixels / inch14,15. This software will quantify the fluorescence emitted from green (wavelength of approximately 510 nm) to red (wavelength of approximately 680 nm), and will assign a numerical value of 0 to 3, which corresponds to the severity of the injury according to the manufacturer's instructions.
photography | 6 MONTHS
  Photography. To standardize photographic conditions, the camera will always be placed at the same distance from the tooth surface. To exclude the influence of moisture on the tooth color, the tooth surfaces will be dried with compressed air for 30s. Clinical photographs will be taken with a digital camera (EOS 5d Mark II camera; Canon, Tokyo, Japan), macro lenses (SP AF100 mm F ⁄ 2.8 Di 1: 1 Macro lenses; Canon, Tokyo, Japan) and flash (MT Twinlight 24- EX; Canon). The camera settings will be as follows: shutter speed 1 ⁄ 125, F29, ISO 200 and automatic white balance. The photographic evaluation will be carried out by the same examiner; Photographs will be randomly designated to avoid measurement bias and will be measured using the L * a * b * scoring method of the Commission Internationale de l'E 'clairage.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain